CLINICAL TRIAL: NCT02807597
Title: Evaluation of LS301 Uptake in Tumors of Patients Undergoing Partial Mastectomy and Sentinel Lymph Node Biopsy for Breast Cancer
Brief Title: Real-time Intraoperative Breast Cancer Visualization for Margin Assessment
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Before LS301's licensing and reformulation, 9 patients received LS301-HSA (Phase 1a) , but since no patients were recruited (in Phase 1b) before the product expired, this study has been terminated.
Sponsor: Samuel Achilefu (Other)
Responsible Party: Sponsor-Investigator, Samuel Achilefu, Professor & Chair, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2022-0385
Record Dates: First submitted 2016-06-13; First posted 2016-06-21 (Estimated); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: A rolling six design will be used to enroll patients in the phase I dose escalating portion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (5):
- Phase I Dose Level 1: LS301 (Experimental): * Patient will undergo surgery 4-24 hours after administration of LS301 (0.05 mg/kg)
  * Excised tissue will be examined for the presence of LS301 fluorescence using the Cancer Vision Goggles (CVG) to determine if LS301 accumulated in the breast cancer. The investigators will quantify fluorescence intensity in the cancer to establish the feasibility of observing LS301 fluorescence with the imaging system. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.
  Interventions: Drug: LS301; Device: Cancer Vision Goggles and standard fluorescence imaging systems; Procedure: Surgery
- Phase I Dose Level 2: LS301 (Experimental): * Patient will undergo surgery 4-24 hours after administration of LS301 (0.075 mg/kg)
  * Excised tissue will be examined for the presence of LS301 fluorescence using the Cancer Vision Goggles (CVG) to determine if LS301 accumulated in the breast cancer. The investigators will quantify fluorescence intensity in the cancer to establish the feasibility of observing LS301 fluorescence with the imaging system. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.
  Interventions: Drug: LS301; Device: Cancer Vision Goggles and standard fluorescence imaging systems; Procedure: Surgery
- Phase I Dose Level 3: LS301 (Experimental): * Patient will undergo surgery 4-24 hours after administration of LS301 (0.1 mg/kg)
  * Excised tissue will be examined for the presence of LS301 fluorescence using the Cancer Vision Goggles (CVG) to determine if LS301 accumulated in the breast cancer. The investigators will quantify fluorescence intensity in the cancer to establish the feasibility of observing LS301 fluorescence with the imaging system. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.
  Interventions: Drug: LS301; Device: Cancer Vision Goggles and standard fluorescence imaging systems; Procedure: Surgery
- Phase I Dose Expansion: LS301 (Experimental): * Patient will undergo surgery 4-24 hours after administration of LS301 (dose to be determined in Phase I dose escalation portion)
  * 9 patients will be enrolled (6 invasive ductal carcinoma and 3 DCIS)
  * Excised tissue will be examined for the presence of LS301 fluorescence using the Cancer Vision Goggles (CVG) to determine if LS301 accumulated in the breast cancer. The investigators will quantify fluorescence intensity in the cancer to establish the feasibility of observing LS301 fluorescence with the imaging system. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.
  Interventions: Drug: LS301; Device: Cancer Vision Goggles and standard fluorescence imaging systems; Procedure: Surgery
- Phase II: LS301 (Experimental): * Patient will undergo surgery 4-24 hours after administration of LS301 (dose to be determined in Phase I portion)
  * Excised tissue will be examined for the presence of LS301 fluorescence using the Cancer Vision Goggles (CVG) to determine if LS301 accumulated in the breast cancer. The investigators will quantify fluorescence intensity in the cancer to establish the feasibility of observing LS301 fluorescence with the imaging system. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.
  Interventions: Drug: LS301; Device: Cancer Vision Goggles and standard fluorescence imaging systems; Procedure: Surgery

INTERVENTIONS:
Drug: LS301 — -LS301 is a small molecule consisting of a NIR fluorescent dye and an octapeptide that is cyclized through a disulfide bond.
Device: Cancer Vision Goggles and standard fluorescence imaging systems — -Member of the operating team will wear the CVG during surgery
  Other Names: CVG
Procedure: Surgery — -Standard of care

SUMMARY:
The investigators' preclinical data have demonstrated the feasibility of fluorescence-guided tumor resection by Cancer Vision Goggles (CVG) with LS301 in animal models. In this study, the investigators will conduct intraoperative imaging procedures that have minimal interference with ongoing surgery. The underlying hypothesis is that the accurate detection of all cancer cells highlighted by LS301 during surgery will reduce the number of breast cancer patients with margin positivity to less than 5%, compared to the current surgical paradigm of greater than 20%. The pilot study will obtain critical data required to address the larger question of surgical margin assessment in a full Phase I clinical trial.

Phase 1: to determine the safety and optimal imaging dose of LS301 injected in breast cancer patients.

Phase 2: to determine the ability of this novel fluorescence imaging agent to predict the presence of positive margins around partial mastectomy specimens and positive SLNs during surgical therapy for breast cancer.

DETAILED DESCRIPTION:
A rolling six design which is intended for relatively safe trials and shortening the study duration is proposed for the phase 1 portion 74. In the rolling six design, three to six patients can be enrolled to a dose each time. The dose de-escalation occurs when two or more DLT occur at a dose level while dose escalation occurs when 3/3, 4/4, 5/5, 5/6 or 6/6 patients are evaluated without DLT 75. Three dose levels will be tested in the phase I study, 0.05, 0.075 and 0.10 mg/kg. LS301 will be administered intravenously at a starting dose of 0.05 mg/kg to a cohort of six patients and escalate/de-escalate following the decision rule of the rolling six design. Once six patients have been included at the current dose level, inclusions are suspended until at least five of the six patients have completed the procedure without DLT observed in the evaluation period. MTD is hit where two or more patients out of six at a dose level experience DLT. The investigators do not expect any serious adverse events related to LS301 at the initial Dose Level 1. Once the MTD is determined, an expansion cohort with 9 patients will be tested at the MTD and an optimal imaging dose will be recommended for the subsequent phase II trial.

At the completion of the expansion cohort, a single arm phase 2 trial will be performed at the optimal imaging dose. A breast surgeon will perform breast conserving surgery per standard of care. At the completion of the surgery, a second investigator (to reduce bias in data collection) will wear the cancer vision goggle (CVG) to visualize the excised tissue to determine if there are any positive margins based on the presence of LS301 fluorescence. If any positive margins are observed, the subject will be considered to have a positive margin; otherwise, the margin is considered negative. The excised tissue will later be examined by a breast cancer pathologist. Standard pathologic techniques will be used to determine if there are positive margins. Particular attention will be paid to the sites marked following CVG assessment to confirm whether the margin is positive or negative at any of these sites, or positive at other locations not identified by CVG. No interventions will be allowed based on the CVG results.

This study was initiated at Washington University in St. Louis and is being transferred to UTSW. Phase 1a was initiated at Washington University in St. Louis where 9 subjects were enrolled. The PI is continuing with Phase 1B at UTSW where 9 more subjects will be enrolled. Once completed, the results of Phase 1 (a and b) will be sent to the FDA for review. Phase II will begin once the FDA has reviewed the interim data and authorized Phase II to open. After phase 1 data has been submitted to and discussed with the FDA, an additional cohort of 88 patients will be enrolled to the phase 2 portion of the trial to assess the diagnostic capabilities of LS301 for identification of positive margins at surgery. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Stage I-II breast cancer patients undergoing breast-conserving therapy and SLN biopsy.
* Negative nodal basin clinical exam.
* At least 18 years of age.
* Able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Contraindications for surgery.
* Receiving any investigational agents.
* History of allergic reactions attributed to ICG or other agents used in the study, include known iodide or seafood allergy. The investigators do not expect many of these adverse reactions with LS301 because it is not radioactive and does not possess iodinated counter ions.
* Presence of underlying lung disease
* Pregnant. Female patients of childbearing potential must have a negative serum or urine pregnancy test no more than 7 days before start of participation.
* Breastfeeding. Patients who are breastfeeding are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LS301.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Achilefu, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center; Deborah Farr, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 subjects started and completed phase 1a period (14-15 months). Study was terminated and did not proceed to the next phases planned in the next period 2.
Groups:
- Phase I Dose Level 1: LS301: * Patient will undergo surgery 4-24 hours after administration of LS301 (0.05 mg/kg)
  * Excised tissue will be examined for the presence of LS301 fluorescence using the Cancer Vision Goggles (CVG) to determine if LS301 accumulated in the breast cancer. The investigators will quantify fluorescence intensity in the cancer to establish the feasibility of observing LS301 fluorescence with the imaging system. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.
  LS301: -LS301 is a small molecule consisting of a NIR fluorescent dye and an octapeptide that is cyclized through a disulfide bond.
  Cancer Vision Goggles and standard fluorescence imaging systems: -Member of the operating team will wear the CVG during surgery
  Surgery: -Standard of care
- Phase I Dose Level 2: LS301: * Patient will undergo surgery 4-24 hours after administration of LS301 (0.075 mg/kg)
  * Excised tissue will be examined for the presence of LS301 fluorescence using the Cancer Vision Goggles (CVG) to determine if LS301 accumulated in the breast cancer. The investigators will quantify fluorescence intensity in the cancer to establish the feasibility of observing LS301 fluorescence with the imaging system. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.
  LS301: -LS301 is a small molecule consisting of a NIR fluorescent dye and an octapeptide that is cyclized through a disulfide bond.
  Cancer Vision Goggles and standard fluorescence imaging systems: -Member of the operating team will wear the CVG during surgery
  Surgery: -Standard of care
- Phase I Dose Level 3: LS301: * Patient will undergo surgery 4-24 hours after administration of LS301 (0.1 mg/kg)
  * Excised tissue will be examined for the presence of LS301 fluorescence using the Cancer Vision Goggles (CVG) to determine if LS301 accumulated in the breast cancer. The investigators will quantify fluorescence intensity in the cancer to establish the feasibility of observing LS301 fluorescence with the imaging system. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.
  LS301: -LS301 is a small molecule consisting of a NIR fluorescent dye and an octapeptide that is cyclized through a disulfide bond.
  Cancer Vision Goggles and standard fluorescence imaging systems: -Member of the operating team will wear the CVG during surgery
  Surgery: -Standard of care
- Phase I Dose Expansion: LS301: * Patient will undergo surgery 4-24 hours after administration of LS301 (dose to be determined in Phase I dose escalation portion)
  * 9 patients will be enrolled (6 invasive ductal carcinoma and 3 DCIS)
  * Excised tissue will be examined for the presence of LS301 fluorescence using the Cancer Vision Goggles (CVG) to determine if LS301 accumulated in the breast cancer. The investigators will quantify fluorescence intensity in the cancer to establish the feasibility of observing LS301 fluorescence with the imaging system. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.
  LS301: -LS301 is a small molecule consisting of a NIR fluorescent dye and an octapeptide that is cyclized through a disulfide bond.
  Cancer Vision Goggles and standard fluorescence imaging systems: -Member of the operating team will wear the CVG during surgery
  Surgery: -Standard of care
- Phase II: LS301: * Patient will undergo surgery 4-24 hours after administration of LS301 (dose to be determined in Phase I portion)
  * Excised tissue will be examined for the presence of LS301 fluorescence using the Cancer Vision Goggles (CVG) to determine if LS301 accumulated in the breast cancer. The investigators will quantify fluorescence intensity in the cancer to establish the feasibility of observing LS301 fluorescence with the imaging system. FDA-approved fluorescence imaging systems may be used to benchmark CVG data.
  LS301: -LS301 is a small molecule consisting of a NIR fluorescent dye and an octapeptide that is cyclized through a disulfide bond.
  Cancer Vision Goggles and standard fluorescence imaging systems: -Member of the operating team will wear the CVG during surgery
  Surgery: -Standard of care
Period: Phase 1 Period (14-15 Months)
Arm/Group | Phase I Dose Level 1: LS301 | Phase I Dose Level 2: LS301 | Phase I Dose Level 3: LS301 | Phase I Dose Expansion: LS301 | Phase II: LS301
Started | 3 | 3 | 3 | 0 | 0
Completed | 3 | 3 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase 2 Period (2 Months)
Arm/Group | Phase I Dose Level 1: LS301 | Phase I Dose Level 2: LS301 | Phase I Dose Level 3: LS301 | Phase I Dose Expansion: LS301 | Phase II: LS301
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data collected is only from Subjects who were enrolled at WashU for phase 1a. No subjects were enrolled after that for rest of the phases and the study was terminated.
Groups:
- LS301 (0.05 mg/Kg): Subjects who were enrolled for LS301 dose (0.05 mg/Kg) in Phase 1a. Phase 1b and rest of the phases did not start.
- LS301 (0.075 mg/Kg): Subjects who were enrolled for LS301 dose (0.075 mg/Kg) in Phase 1a. Phase 1b and rest of the phases did not start.
- LS301 (0.1 mg/Kg): Subjects who were enrolled for LS301 dose (0.1 mg/Kg) in Phase 1a. Phase 1b and rest of the phases did not start.
- Total: Total of all reporting groups
Arm/Group | LS301 (0.05 mg/Kg) | LS301 (0.075 mg/Kg) | LS301 (0.1 mg/Kg) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Customized [Count of Participants; unit: Participants]
  54 to 74 years | 3 | 3 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 9
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 3 | 9
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 27.17 (0.49) | 30.9 (6.14) | 27.17 (3.38) | 28.41 (3.98)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Related Adverse Events of LS301 in Breast (Phase I)
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Time Frame: Time of injection to 3 hours post-injection
Population: Since this outcome measure is specific to phase I, no data was collected for Phase I Dose Expansion Arm and Phase II Arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1: LS301 | Phase I Dose Level 2: LS301 | Phase I Dose Level 3: LS301 | Phase I Dose Expansion: LS301 | Phase II: LS301
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Receiving Optimal Imaging Dose of LS301 (Phase I)
Description: * Optimal dose will be the dose at which fewer than 2 dose-limiting toxicities (DLTs) are observed and optimal image quality is observed. It need not be the maximum tolerated dose (MTD) if optimal image quality is observed at a lower dose than the MTD.
  * DLT is defined as any grade 2 or above toxicity that occurs during the hour after injection that is considered possibly, probably, or definitely related to LS301
  * Toxicities will be graded using the NCI Common Terminology Criteria for Adverse Events version 5.0
Time Frame: 14-15 months
Population: This outcome is specific to Phase 1 and since due to study termination, it never proceeded to the next phases after phase 1a was completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1: LS301 | Phase I Dose Level 2: LS301 | Phase I Dose Level 3: LS301 | Phase I Dose Expansion: LS301 | Phase II: LS301
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Ability of LS301 to Predict Presence of Positive Margins Around Partial Mastectomy (Phase II)
Description: -The histopathological results of margin positivity has the following possible results: margin negative, margin positive at LS301 and CVG identified locations, margin positive at LS301 and CVG unidentified locations. Using LS301 and CVG, the exercised tissue will be considered to be margin positive and have ink marked at the identified locations if any positive margins are observed; otherwise, the margin is considered negative. Diagnostic test characteristics (sensitivity and specificity) of LS301 and CVG for margin positivity by histology will established and margin positivity rate, defined as the proportion of tumors with histopathologically confirmed positive margins but missed by CVG, will be estimated.
Time Frame: Day 1 (at the time of surgery)
Population: Data not collected for this outcome specific for phase II since study was terminated and did not proceed beyond phase 1a.
Arm/Group | Phase I Dose Level 1: LS301 | Phase I Dose Level 2: LS301 | Phase I Dose Level 3: LS301 | Phase I Dose Expansion: LS301 | Phase II: LS301
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Toxicity of LS301 in Breast as Measured by Related Adverse Events (Phase II)
Description: as for outcome 1
Time Frame: up to 48 hours post LS301 injection
Population: as for outcome 3
Arm/Group | Phase I Dose Level 1: LS301 | Phase I Dose Level 2: LS301 | Phase I Dose Level 3: LS301 | Phase I Dose Expansion: LS301 | Phase II: LS301
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 14-15 months
Description: 9 subjects started and completed phase 1a period (14-15 months). Study was terminated and did not proceed to the next phases (phase 1b and phase 2) planned in the next period 2.
Arm/Group | Phase I Dose Level 1: LS301 | Phase I Dose Level 2: LS301 | Phase I Dose Level 3: LS301 | Phase I Dose Expansion: LS301 | Phase II: LS301
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Before LS301's licensing and reformulation, 9 patients received LS301-HSA (Phase 1a) , but since no patients were recruited (in Phase 1b) before the product expired, this study has been terminated. Therefore, no data was collected and reported for phase 1b and phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT02807597/Prot_SAP_002.pdf
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT02807597/ICF_003.pdf